## Perioperative Oral Steroids for Chronic Rhinosinusitis Without Polyps

Statistical Analysis Plan

NCT02748070

July 2, 2020

Julia Noel, Principal Investigator Stanford University Stanford, California 94305

The planned sample size was 75 patients. By power analysis, we required 50 patients to achieve statistical significance. We collected outcome measures of SNOT-22 and Lund-Kennedy endoscopy scores at the following time points: preoperative baseline, and postoperatively at 1 week, 1 month, 3 months, and 6 months.

All statistical analyses were performed using Stata 15 (Stata Statistical Software: Release 15; StataCorp LP, College Station, Texas). SNOT-22 total scores, SNOT-22 subdomain scores, Lund-Kennedy endoscopic scores, and adverse effects were compared between prednisone and placebo groups at each time point using t-tests.